CLINICAL TRIAL: NCT02377518
Title: Quantitative Ventilation Imaging With Dual Energy Computed Tomography
Brief Title: DECT Ventilation Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of device used for dual energy computed tomography with Xenon
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5601
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: For Oncologic Patients; Potentially Operable Lung Tumor; With a Recent (Less Than 1 Month) VQ Scan; For Lung Transplant Recipients; Single of Bilateral Lung Transplant; From 5 Months Onwards; With Recent (Less Than 1 Month) Respiratory Functional Explorations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oncologic patients (Experimental): Prediction of postoperative pulmonary function.
  Patients with an operable lung cancer: dual energy computed tomography with Krypton will be tested to estimate the postoperative FEV1
  Interventions: Radiation: Single source dual energy compted tomography (CT750HD, General Electric, USA) with Krypton as a gaseous contrast media
- lung transplant recipients (Experimental): Detection of BOS
  6 months+ lung transplant recipients will be tested using dual energy computed tomography with Krypton, with acquisition in the end-inspiratory and end-expiratory phase, in search of regional air trapping.
  Interventions: Radiation: Single source dual energy compted tomography (CT750HD, General Electric, USA) with Krypton as a gaseous contrast media

INTERVENTIONS:
Radiation: Single source dual energy compted tomography (CT750HD, General Electric, USA) with Krypton as a gaseous contrast media

SUMMARY:
Demonstrate the feasibility of dual energy computed tomography using Krypton as a gaseous contrast media in order to study the in vivo ventilation.

Two different clinical situations will be tested :

* Prediction of postoperative pulmonary function for oncologic patients
* Detection of Bronchiolitis Obliterans in lung transplant recipients.

ELIGIBILITY:
Inclusion criteria:

For oncologic patients :

* Potentially operable lung tumor
* With a recent (less than 1 month) V/Q scan

For lung transplant recipients :

* Single of bilateral lung transplant
* From 5 months onwards
* With recent (less than 1 month) respiratory functional explorations

Exclusion criteria:

* Impossibility to follow simple orders or control one's respiration
* Known Krypton hypersensitivity
* History of malignant hyperthermia
* Increased intracranial pressure
* Minors
* Pregnant Women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Image quality on a qualitative 5 levels scale | 1 day of DECT ventilation imaging

SECONDARY OUTCOMES:
Radiation dose | 1 day of DECT ventilation imaging
Image noise with measurement of signal to noise and contrast to noise ratios | 1 day of DECT ventilation imaging
Total examination time | 1 day of DECT ventilation imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie B - Nouvel Hôpital Civil - CHRU de Strasbourg, Strasbourg, France